CLINICAL TRIAL: NCT02198482
Title: Dose Finding Safety Run-in Phase Followed by a Randomized Phase II Trial of Intensive Chemotherapy With or Without Volasertib (BI 6727) Administered Prior or After Chemotherapy in Patients With Newly Diagnosed High-Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML)
Brief Title: Trial of Intensive Chemotherapy With or Without Volasertib in Patients With Newly Diagnosed High-Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: development program of study drug volasertib was stopped by Boehringer Ingelheim due to manufacturing problems
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 20-13; 2014-000477-39 (EudraCT Number)
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Acute Myeloid Leukemia (AML); High-risk Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia (AML); Volasertib; High-risk Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 6727; Cytarabine; Daunorubicin; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Daunorubicin, Cytarabine (DA) (Active Comparator): DA
  Induction I:
  * Daunorubicin 60 mg/m² i.v., d 1-3
  * Cytarabine 100 mg/m² cont. i.v., d 1-7
  Induction II:
  * Daunorubicin 50 mg/m² i.v. d 1-3
  * Cytarabine 100 mg/m² cont. i.v., d 1-5
  Consolidation therapy:
  Patients with genetic favourable risk and those patients not eligible for allogeneic HSCT due to comorbidities, high HCT-CI or patient wish will proceed to 3 cycles of age-adapted consolidation therapy with mitoxantrone and intermediate-dose cytarabine (MiDAC).
  * Mitoxantrone Younger adults (18 to 60 yrs): 10 mg/m2 by i.v. on day 1. Elderly patients (>60 yrs): 8 mg/m2 by i.v. infusion on day 1.
  * Intermediate-dose cytarabine:
  Younger adults (18 to 60 yrs): 1500 mg/m2 q12h on days 1-3 Elderly patients (>60 yrs): 1000 mg/m2 q12h on days 1-3 An allogeneic HSCT is intended for patients with intermediate I/II and adverse-risk genetics. Optionally, one cycle of consolidation with MiDAC may be given prior to alloHSCT.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Mitoxantrone
- Volasertib, Daunorubicin, Cytarabine (Experimental): VDA
  Induction I
  * Volasertib i.v., d1
  * Daunorubicin 60 mg/m² i.v., d 2-4
  * Cytarabine 100 mg/m² cont. i.v., d 2-8 Induction II
  * Volasertib i.v., d1
  * Daunorubicin 50 mg/m² i.v. d 2-4
  * Cytarabine 100 mg/m² cont. i.v., d 2-6
  Consolidation therapy:
  Patients with genetic favourable risk and those patients not eligible for allogeneic HSCT will proceed to 3 cycles of age-adapted consolidation therapy with mitoxantrone and intermediate-dose cytarabine in combination with Volasertib (V-MiDAC).
  * Volasertib i.v., d1
  * Mitoxantrone Younger adults (18 to 60 yrs): 10 mg/m2 by i.v. on day 2. Elderly patients (>60 yrs): 8 mg/m2 by i.v. on day 2.
  * Intermediate-dose cytarabine:
  Younger adults (18 to 60 yrs): 1500 mg/m2 q12h on days 2-4 Elderly patients (>60 yrs): 1000 mg/m2 q12h on days 2-4 An allogeneic HSCT is intended for patients with intermediate I/II and adverse-risk genetics. Optionally, one cycle of consolidation with V-MiDAC may be given prior to alloHSCT.
  Interventions: Drug: Volasertib; Drug: Cytarabine; Drug: Daunorubicin; Drug: Mitoxantrone
- Daunorubicin, Cytarabine, Volasertib (Experimental): DAV
  Induction I
  * Volasertib i.v., d7
  * Daunorubicin 60 mg/m² i.v., d 1-3
  * Cytarabine 100 mg/m² i.v., d 1-7 Induction II
  * Volasertib i.v., d5
  * Daunorubicin 50 mg/m² i.v. d 1-3
  * Cytarabine 100 mg/m² cont. i.v., d 1-5
  Consolidation therapy:
  Patients with genetic fav. risk and those patients not eligible for alloHSCT will proceed to 3 cycles of age-adapted consolidation therapy with mitoxantrone and intermediate-dose cytarabine in combination with Volasertib (MiDAC-V).
  * Volasertib i.v., d4
  * Mitoxantrone Younger adults (18 to 60 yrs): 10 mg/m2 by i.v. on day 1. Elderly patients (>60 yrs): 8 mg/m2 by i.v. on day 1.
  * Intermediate-dose cytarabine:
  Younger adults (18 to 60 yrs): 1500 mg/m2 q12h on days 1-3 Elderly patients (>60 yrs): 1000 mg/m2 q12h on days 1-3 An allogeneic HSCT is intended for patients with intermediate I/II and adverse-risk genetics. Optionally, one cycle of consolidation with MiDAC-V may be given prior to alloHSCT.
  Interventions: Drug: Volasertib; Drug: Cytarabine; Drug: Daunorubicin; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Volasertib
  Arms: Daunorubicin, Cytarabine, Volasertib; Volasertib, Daunorubicin, Cytarabine
Drug: Cytarabine
  Other Names: ARA-cell
Drug: Daunorubicin
  Other Names: Daunoplastin
Drug: Mitoxantrone
  Other Names: Novantron

SUMMARY:
Randomized Phase II Trial of Intensive Chemotherapy With or Without Volasertib (BI 6727) in Patients With Newly Diagnosed High-Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML)

DETAILED DESCRIPTION:
The trial is a randomized, Phase II, open label multi-center trial in adult patients with newly diagnosed AML or high-risk MDS as defined in the inclusion/exclusion criteria.

An initial safety run-in study will be performed administering intensive induction therapy consisting of daunorubicin and cytarabine with the study drug volasertib administered prior or after chemotherapy, as well as consolidation therapy consisting of intermediate-dose cytarabine with the study drug volasertib administered prior or after chemotherapy. After establishing the volasertib dose, the randomized Phase II portion of the trial will begin:

Patients will be equally randomized to DA (daunorubicin, cytarabine), V-DA (volasertib administered prior to daunorubicin, cytarabine), and DA-V (volasertib administered after daunorubicin, cytarabine). All patients will receive a second induction cycle with reduced daunorubicin and cytarabine doses. Patients refractory to the first induction cycle and patients not achieving a CR/CRi after two induction cycles will be off-study and followed up.

Patients in CR/CRi after induction therapy will proceed to consolidation therapy. Consolidation will be stratified based on the genetic risk profile (according to ELN criteria) and patient-related factors (e.g., age, HCT-CI, comorbidities, patient wish). Patients with a favorable genetic risk profile and those patients considered ineligible for allogeneic HCT will receive repetitive cycles of consolidation according to initial randomization, either MiDAC, V-MiDAC (volasertib administered prior to cytarabine), or MiDAC-V (volasertib administered after cytarabine). All other patients are assigned to allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of acute myeloid leukemia (AML) or related precursor neoplasm, or acute leukemia of ambiguous lineage according to the current World Health Organization (WHO) classification, or patients with myelodysplastic syndrome (MDS) classified as refractory anemia with excess blasts-2 (RAEB-2)
* Consent for a genetic assessment in AMLSG central laboratory
* Patients considered eligible for intensive chemotherapy
* ECOG performance status of ≤ 2
* Age >= 18; there is no upper age limit
* No prior chemotherapy for acute leukemia except hydroxyurea for up to 5 days during the diagnostic screening phase; patients may have received prior therapy for myelodysplastic syndrome.
* Non-pregnant and non-nursing. Due to the teratogenic potential of volasertib in humans, pregnant or nursing patients may not be enrolled. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control - one highly effective method (e.g., IUD, hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (e.g., latex condom, diaphragm, or cervical cap) for 6 months after therapy is stopped. "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
* Men must agree not to father a child and must use a latex condom during any sexual contact with women of childbearing potential while receiving therapy and for 6 months after therapy is stopped, even if they have undergone a successful vasectomy
* Signed written informed consent

Exclusion Criteria:

* Patients with acute promyelocytic leukemia exhibiting t(15;17)(q22;q12); PML-RARA, or with variant translocations
* Prior treatment with volasertib or any other PLK1 inhibitor
* Performance status WHO >2 (see Appendix I)
* Patients with ejection fraction <50% by echocardiography within 14 days of day 1
* QTcF prolongation >470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome). The QTcF will be calculated as the mean of 3 ECGs taken at screening.
* Any clinically significant, advanced or unstable disease or history of that may interfere with primary or secondary variable evaluations or put the patient at special risk, such as:

  * creatinine >1.5x upper normal serum level;
  * total bilirubin, AST or AP >2.5x upper normal serum level;
  * heart failure NYHA III/IV,
  * uncontrolled hypertension,
  * unstable angina,
  * serious cardiac arrhythmia;
  * severe obstructive or restrictive ventilation disorder
  * uncontrolled infection
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Known or suspected active alcohol or drug abuse
* Known positive for HIV, active HBV, HCV, or hepatitis A infection
* Hematologic disorder independent of leukemia
* No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation.
* No consent for biobanking.
* Current participation in any other interventional clinical study within 30 days before the first administration of the investigational product or at any time during the study
* Breast feeding women or women with a positive pregnancy test at Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission (CR) and CR with incomplete blood count recovery (CRi) | 2 months

SECONDARY OUTCOMES:
Cumulative incidence of relapse | 4 years
Cumulative incidence of death | 4 years
Relapse-free survival | 4 years
Event-free survival | 4 years
Overall survival | 4 years
Incidence and intensity of adverse events | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Döhner, Prof. Dr., Principal Investigator — AMLSG Clinical Trials Office; Peter Paschka, MD, Study Chair — University Hospital Ulm
Locations (45):
- Germany (45):
  - Hospital Aschaffenburg, Aschaffenburg
  - Helios Hospital Bad Saarow, Bad Saarow
  - Vivantes Hospital Am Urban, Berlin
  - Vivantes Hospital Neukölln, Berlin
  - Charite Berlin Campus Virchow Hospital, Berlin
  - Knappschaftskrankenhaus Bochum-Langendeer, Bochum
  - University Hospital Bonn, Bonn
  - Community Hospital Braunschweig, Braunschweig
  - Hospital Darmstadt, Darmstadt
  - University Hospital Düsseldorf, Düsseldorf
  - Hospital Essen, Protestant Hospital Essen-Werden, Essen
  - Hospital Esslingen, Esslingen am Neckar
  - Malteser Hospital St. Franziskus, Flensburg
  - Hospital Frankfurt-Höchst, Frankfurt
  - Medical Care Unit Osthessen, Fulda
  - University Hospital Gießen, Giessen
  - Wilhelm-Anton-Hospital Goch, Goch
  - University Hospital Göttingen, Göttingen
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Asklepios Hospital Altona, Hamburg
  - Hospital Hanau, Hanau
  - KRH Hospital Siloah-Oststadt-Heidehaus, Hanover
  - Hannover Medical School, Hanover
  - SLK-Hospital Heilbronn, Heilbronn
  - Marienhospital Herne, Herne
  - University Hospital des Saarlandes, Homburg/Saar
  - Community Hospital Karlsruhe, Karlsruhe
  - University Hospital Schleswig-Holstein, Kiel
  - Caritas Hospital Lebach, Lebach
  - Hospital Lippe-Lemgo, Lemgo
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Johannes Gutenberg Mainz, Mainz
  - Johannes Wesling Hospital Minden, Minden
  - Stauferklinikum Schwäbisch-Gmünd, Mutlangen
  - Hospital Schwabing, München
  - Hospital rechts der Isar München, München
  - Hospital Oldenburg, Oldenburg
  - Hospital Passau, Passau
  - Hospital Stuttgart, Stuttgart
  - Diakonie Hospital Stuttgart, Stuttgart
  - Hospital Traunstein, Traunstein
  - Mutterhaus der Borromäerinnen, Trier
  - Hospital Barmherzige Brüder Trier, Trier
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm